CLINICAL TRIAL: NCT06883838
Title: Enhancing Primary Care Capacity for Cancer Survivorship Care Delivery in Community Health Clinics
Brief Title: Project CASCADE: Community and Academic Synergy for Cancer Survivorship Care Delivery Enhancement
Acronym: CASCADE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Bijal.A.Balasubramanian, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HSC-SPH-24-0777; U01CA290663 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivorship
Keywords: cancer survivorship; community health centers; care delivery; primary care

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial (SW-CRT). There will be 4 clusters (CHCs) having 2 practices each.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Step 1 (2 clinics)-6 months control then 12 months intervention (Experimental)
  Interventions: Behavioral: Survivorship care delivery intervention
- Step 2 (2 clinics)-12 months control then 12 months intervention (Experimental)
  Interventions: Behavioral: Survivorship care delivery intervention
- Step 3 (2 clinics)-18 months control then 12 months intervention (Experimental)
  Interventions: Behavioral: Survivorship care delivery intervention
- Step 4 (2 clinics)- 24 months control then 12 months intervention (Experimental)
  Interventions: Behavioral: Survivorship care delivery intervention

INTERVENTIONS:
Behavioral: Survivorship care delivery intervention — Guided by the Practical, Robust Implementation and Sustainability Model (PRISM), the intervention includes three evidence-based components:
  1. Training: This will include provider-to-provider tele-mentoring using Enhancing Community Health Outcomes (ECHO).
  2. Tracking: This includes systematically assessing cancer history and monitoring survivors' care to plan and organize subsequent care.
  3. Coordinating care for cancer survivors. Each clinic leader will designate a staff member (or members) as the care coordinator champion after exploring current clinic staff, skills, and capacity of various staff roles.

SUMMARY:
The purpose of this study is to implement a clinic-level cancer survivorship care delivery intervention in partnership with community health center clinicians, patients, and community representatives to test effectiveness of the intervention to improve patient and clinician outcomes and to evaluate implementation of the intervention using an iterative, concurrent mixed-methods approach guided by the Practice Change Model.

ELIGIBILITY:
Inclusion Criteria (participants):

-at least one visit to the Community Health Centers (CHCs) in the prior year

Exclusion Criteria (participants):

- no history of cancer recorded in the problem list or past medical history in the medical record

Inclusion Criteria (clinicians):

-employed clinicians (e.g. physicians, nurses, pharmacists, or other allied health professionals) and non-clinician staff of the participating CHC clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5584 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible cancer survivors screened for second primary cancers | every 6 months from baseline to end of study (about 36 months from baseline)
  Data derived from electronic health records

SECONDARY OUTCOMES:
Change in proportion of primary care clinician knowledge of cancer survivorship care | baseline, six months following end of intervention period
  Assessed by self-administered survey
Change proportion of survivors that report better experience of provider communication as assessed by the adapted Consumer Assessment of Healthcare Providers and Systems (CAHPS 4.0) | baseline, six months following end of intervention period
Change proportion of survivors that report better experience of care coordination as assessed by the adapted Consumer Assessment of Healthcare Providers and Systems (CAHPS 4.0) | baseline, six months following end of intervention period
Proportion of survivors who received guideline-recommended surveillance for the most prevalent cancers (breast colorectal, prostate, cervical, and lung) | every 6 months from baseline to end of study (about 36 months from baseline)
  Per national guidelines [National Comprehensive Cancer Network (NCCN), U.S. Preventive Services Task Force (USPSTF)]; data derived from electronic health records

CONTACTS AND LOCATIONS:
Overall Officials: Bijal Balasubramanian, MBBS, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Simon Craddock Lee, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Texas Health Science Center, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No